CLINICAL TRIAL: NCT04642404
Title: Cannabidiol (CBD) for the Management of Emergency Dental Pain
Brief Title: CBD for Dental Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20200305H
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Odontalgia; Toothache
Keywords: Cannabidiol (CBD); Opioid; Dose; Dental; Pain; Epidiolex; CBD
MeSH Terms: conditions — Toothache; Pain | interventions — Cannabidiol; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients who satisfy eligibility criteria and provide written informed consent will be randomly assigned to either 1) CBD 10mg/kg single dose (drug: Epidiolex 100mg/ml solution) or 2) CBD 20mg/kg single dose, or 3) Placebo group (drug: placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Epidiolex 10mg/kg single dose (Experimental): After drug administration, subjects will be monitored for 3 hours, and pain intensity and safety data will be collected at various time points. Ibuprofen 600mg (or acetaminophen/codeine 650/60mg, if a contraindication for ibuprofen exists) will be provided in the 3-hour observation period as rescue medication if needed. Subjects will be encouraged to wait at least 60min after administration of the drug study before consuming the rescue medication. It will be given at the patient's request. If rescue medication was required, the study drug will still be dosed as per protocol, and time-to -rescue analysis will be performed. Then, the recommended root canal therapy will be performed the same or the next day.
  Interventions: Drug: Epidiolex 100 mg/mL Oral Solution
- Epidiolex 20mg/kg single dose (Experimental): The 20mg/kg dose is the maximum recommended daily dose from the manufacturer. After drug administration, subjects will be monitored for 3 hours, and pain intensity and safety data will be collected at various time points. Ibuprofen 600mg (or acetaminophen/codeine 650/60mg, if a contraindication for ibuprofen exists) will be provided in the 3-hour observation period as rescue medication if needed. Subjects will be encouraged to wait at least 60min after administration of the drug study before consuming the rescue medication. It will be given at the patient's request. If rescue medication was required, the study drug will still be dosed as per protocol, and time-to -rescue analysis will be performed. Then, the recommended root canal therapy will be performed the same or the next day.
  Interventions: Drug: Epidiolex 100 mg/mL Oral Solution
- Placebo group (Placebo Comparator): Placebo drug will be a solution with the same taste, texture and color as the drug. After drug administration, subjects will be monitored for 3 hours, and pain intensity and safety data will be collected at various time points. Ibuprofen 600mg (or acetaminophen/codeine 650/60mg, if a contraindication for ibuprofen exists) will be provided in the 3-hour observation period as rescue medication if needed. Subjects will be encouraged to wait at least 60min after administration of the drug study before consuming the rescue medication. It will be given at the patient's request. If rescue medication was required, the study drug will still be dosed as per protocol, and time-to -rescue analysis will be performed. Then, the recommended root canal therapy will be performed the same or the next day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epidiolex 100 mg/mL Oral Solution — Cannabidiol (CBD): is the primary non-psychoactive and non-addictive compound in cannabis, has already shown potential in treating pain such as arthritis, neuropathic, cancer and chronic pain
  Other Names: Cannabidiol (CBD)
  Arms: Epidiolex 10mg/kg single dose; Epidiolex 20mg/kg single dose
Drug: Placebo — Placebo drug will be a solution with the same taste, texture and color as the drug.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaulate CBD as a therapeutic approach for dental pain. Eligible subjects presented with emergency dental pain will be give a single dose of Epidiolex (FDA-approved CBD) or placebo and will be monitored for 3 hours for pain symptoms and psychologic effects.

DETAILED DESCRIPTION:
CBD is a non-psychoactive, non-addictive compound of cannabis that has shown analgesic and anti-inflammatory properties. Epidiolex is the only FDA-approved oral CBD solution and will be the drug of choice in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-75 years old, ASA I or II
* permanent tooth with moderate to severe odontogenic pain, i.e. ≥30 on a 100mm VAS,
* clinical pulpal diagnosis of irreversible pulpitis or pulpal necrosis, and periapical diagnosis of symptomatic apical periodontitis
* test negative for recent cannabis use and/or other drugs of abuse including alcohol (urine tests collected at screening visit), and participant
* able to understand the forms (English or Spanish) and provide informed written consent.

Exclusion Criteria:

* ASA Class III or IV
* patients with hepatic impairment
* pregnant or lactating women
* Patients on drugs metabolized by enzymes that also metabolize CBD (e.g. clobazam, diazepam, topiramate, warfarin)
* self-reported prior experience inhaling cannabis (either via smoking or vaporization), use of opioids in the month prior to screening/treatment visit, and/or NSAIDS or acetaminophen 6 hours prior to treatment
* unwilling to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Chrepa, DDS MS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of adult patients 18 to 75 y old, presenting at the UT Health School of Dentistry, San Antonio, Texas, with moderate to severe odontogenic pain, defined as ≥30 mm on a 100-mm visual analog scale (VAS)
Period: Overall Study
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group
Started | 21 | 20 | 23
Completed | 20 | 20 | 21
Not Completed | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.66) | 44.75 (11.61) | 43.1 (16.78) | 44.15 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 11 | 40
  Male | 7 | 4 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4 | 2 | 0 | 6
  Hispanic | 11 | 16 | 16 | 43
  Hispanic/Native | 0 | 0 | 1 | 1
  White | 5 | 2 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 21 | 61
Weight [Mean (Standard Deviation); unit: Kg] | 94.37 (21.04) | 87.71 (22.21) | 92.43 (22.7) | 91.50 (21.98)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (6.42) | 33.32 (6.63) | 32.32 (5.5) | 33.04 (6.18)

OUTCOME MEASURES:

1. Primary Outcome: Intra-group VAS Pain Intensity and Maximum Pain Relief
Description: Patients will report their pain level using a 100mm Visual Analogue Scale at baseline, measured at baseline and 180 minutes. Score is measured on a 100mm scale, scored 0-100, with a lower score indicating less pain.
Time Frame: Baseline to 180 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group
Number analyzed (Participants) | 20 | 20 | 21
score on a scale
  Baseline | 63 [51.5 to 79.5] | 69 [59 to 76.25] | 63 [51.7 to 73.5]
  180 minutes | 21 [1 to 38] | 20 [4.5 to 39.2] | 48 [13 to 58.7]

2. Primary Outcome: Bite Force Measurement
Description: Bite force is measured by biting down on the Bite Fork at various times to measure change in value. The digital bite transducer is a previously validated instrument used to assess changes in the bite forces (N) before and after the intervention.
Time Frame: Baseline, 90 minutes and 180 minutes
Measure: Median (Inter-Quartile Range); unit: Newtons
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group
Number analyzed (Participants) | 20 | 20 | 21
Newtons
  Baseline | 61 [42.5 to 100] | 53 [32.5 to 60] | 54 [32.5 to 74.5]
  90 minutes | 86 [56 to 135] | 59 [35.7 to 78.7] | 66 [44.5 to 73.5]
  180 minutes | 80 [68 to 135] | 66 [43 to 82] | 65 [43 to 87.5]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Included: Psychoactive effects, mood changes, and report other side effects after single dose of Epidiolex
Time Frame: 3 hours and 7 Days
Population: All subjects enrolled, regardless of whether they completed the study. Adverse effects were self reported. Some subjects were lost to follow up for the 7 day self assessment, so did not complete the self assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group
Number analyzed (Participants) | 21 | 20 | 23
Participants
  3 hour | 9 | 6 | 1
  7 day: number analyzed (Participants) | 18 | 18 | 22
  7 day | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were reported at 3 hours and at 7 days
Arm/Group | Epidiolex 10mg/kg Single Dose | Epidiolex 20mg/kg Single Dose | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 10/21 | 10/20 | 5/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidiolex 10mg/kg Single Dose (N=21) | Epidiolex 20mg/kg Single Dose (N=20) | Placebo Group (N=23)
Somnolence (Nervous system disorders) | 3 (4) | 3 (3) | 2 (2)
Sedation (General disorders) | 6 (7) | 3 (3) | 1 (1)
Headache (General disorders) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abnormal behavior (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 4 (8) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 4 (6) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Hot Flashes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Double vision (Eye disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04642404/Prot_SAP_000.pdf